CLINICAL TRIAL: NCT05433129
Title: Non-Invasive Mapping of Cerebral Autoregulation Using Near Infrared Spectroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS25527 (B2022:051); RGPIN-2022-03621 (Other Grant/Funding Number: NSERC DG)
Record Dates: First submitted 2022-06-10; First posted 2022-06-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Autoregulation Mapping
Keywords: Near Infrared Spectroscopy; Cerebral Mapping; Cerebral Autoregulation
MeSH Terms: interventions — Neurovascular Coupling

STUDY DESIGN:
Intervention Model Description: Device optimization and assessment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Block Testing (Other): Perturbations to the system will be investigated through a series of testing (block design separated by baseline rest): A. transient hyperemic response testing via carotid compression methods, B. orthostatic challenge responses (lying-to-sit, sit-to-stand),8 C. vascular chemo-reactivity via fast and slow breathing exercises and D. impact of neurovascular coupling through cognitive/Stroop testing. Work here will establish areas for improvement in real time.
  Interventions: Procedure: Transient hyperemic response; Procedure: Orthostatic challenge; Procedure: Vascular chemo-reactivity; Procedure: Neurovascular coupling

INTERVENTIONS:
Procedure: Transient hyperemic response — The transient hyperemic response will be tested via carotid compression method. This test will consist of 5 carotid compressions lasting 5 seconds each with a 60 seconds interval between each compression to allow normalization of the CBF to precompression levels, and the total time for this block would be 6 minutes. The ipsilateral common carotid artery will be compressed for this method, and the response of the middle cerebral artery (MCA) blood flow velocity will be assessed using transcranial doppler (TCD) probe (EMS-9D, Delica). The carotid compressions will only be accepted when there is no further decrease in blood flow velocity can be achieved and stable conditions remained during the whole period of the compression. Otherwise, the compression will be terminated and repeated again after 60 seconds. Satisfactory compression is typically considered to result in a reduction in MCA velocity of 50%, at a minimum.
Procedure: Orthostatic challenge — The orthostatic challenge response will be evaluated by lying-to-sit and sit-to-stand methods 5 times where sitting and standing positions will be held for 3 minutes each for a total block time of 35 minutes. A baseline in lying position will be collected at the start of the block, then the position will be changed from lying to sit for 3 minutes and then position will be changed to standing for another 3 minutes.
Procedure: Vascular chemo-reactivity — vascular chemo-reactivity will be assessed by varying CO2 concentrations through slow and fast breathing exercises with Capnostream 35 Portable Respiratory Monitor (Medtronic Canada) to monitor EtCO2 through nose clip. The breathing trials will occur two times and each of them will have fast and slow trials along with an interval of normal breathing. First time, the normal, fast and slow breathing trials will be 2.5 minutes long while the second time, these breathing trials will be 1.5 minutes long. The normal respiratory rate for adults is 12 breaths/minute, the target slow respiratory rate will be 5 breaths/minute and fast respiratory rate will be 25 breaths/minute as set by metronome. It has been shown that the EtCO2 has a 10% increase during hypoventilation and almost 50% decrease during hyperventilation compared to normal breathing.
Procedure: Neurovascular coupling — The fourth block will evaluate the neurovascular coupling using Automated Neuropsychological Assessment Metrics (ANAM) General Neuropsychological Screening (GNS) Clinical Toolkit which contains 5 tests explained as follows 1) Standard Continuous Performance test will assess sustained attention, concentration and working memory. 2) Manikin test will assess 3D spatial rotation ability, left-right orientation, problem solving and attention. 3) Pursuit Tracking test will measure the visuo-motor control. 4) Switching test will assess divided attention, mental flexibility, and executive function. 5) Stroop test will assess the processing speed, selective attention, interference, and executive functioning with three trial blocks.

SUMMARY:
The investigators propose to employ advanced multi-channel near non-invasive near infrared spectroscopy (NIRS) system married with entirely non-invasive continuous arterial blood pressure (niABP) monitor to create a new wearable and portable imaging system that derives CA maps of the entire brain with high sampling rates at each point.

The objectives of this project are as follows:

1. To perform in vivo testing and optimization of the device using a block-trial design to evaluate the CA mapping system's performance during various perturbations.
2. To explore the impact of aging and sex on regional disparities in CA in a healthy volunteer population using static recording along with perturbation testing.

DETAILED DESCRIPTION:
Objective 1:

To assess functionality and feasibility of real-time application in humans, in vivo testing will occur on a small population (n=50) of healthy human volunteers. Such work will investigate feasibility of the combination monitoring setup, optimal NIRS channel placement using the adjustable OxyMon NIRS cap, ability for pipelines to extract and analyze signals in real time for continuous derivation of NIRS-based CVR metrics at each channel and functionality of CVR map generation in real-time. Finally, the investigators will investigate perturbations to system through a series of testing (block design separated by baseline rest): A. transient hyperemic response testing via carotid compression methods, B. orthostatic challenge responses (lying-to-sit, sit-to-stand), C. vascular chemo-reactivity via fast and slow breathing exercises and D. impact of neurovascular coupling through cognitive/Stroop testing. Work here will establish areas for improvement in real time. The testing and optimization phase will last 18 months. The addition of single rSO2 channel from commercial NIRS will be used to provide a "gold standard" data stream to compare our results to.

Objective 2:

Current understanding of the aging process and sex on continuously assessed CA, and regional disparities, has been hampered by a lack of high-resolution platform. The investigators will evaluate the impact of both age and sex on CA using the newly developed platform through static CA assessments in 200 healthy volunteers. Within the 1-hour period, volunteers will have their age and sex recorded in a de-identified electronic database, have an hour of non-invasive simultaneous 24 Channel OxyMon NIRS , Finapres NOVA ABP, and single channel commercial NIRS rSO2 recording which is divided into static resting state recording and perturbation testing. This will facilitate the derivation of a normative reference range for CA using the platform along with making the dataset richer. Static resting state assessments will be done over the first half hour and in second half hour, perturbations to system will be investigated through a series of testing separated by baseline rest: A. orthostatic challenge responses (lying-to-sit, sit-to-stand), B. vascular chemo-reactivity via fast and slow breathing exercises and C. impact of neurovascular coupling through Stroop testing. The addition of single rSO2 channel from commercial NIRS will be used to provide a "gold standard" data stream to compare our results to.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (male and female)
* Age > 17

Exclusion Criteria:

* History of neurological illness
* History of systemic vascular
* History of cerebrovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
In Vivo testing and optimization of device during various perturbations | 2 years
  To assess functionality and feasibility of real-time application in humans, in vivo testing will occur on a small population of healthy human volunteers. Such work will investigate feasibility of the combination monitoring setup, optimal NIRS channel placement using the adjustable OxyMon NIRS cap, ability for pipelines to extract, and analyze signals in real time for continuous derivation of NIRS-based CVR metrics at each channel and functionality of CVR map generation in real-time.
Explore impact of aging and sex on regional disparities in Cerebral Autoregulation | 3 years
  Current understanding of the aging process and sex on continuously assessed CA, and regional disparities, has been hampered by a lack of high-resolution platform. We will evaluate the impact of both age, and sex on CA using the newly developed platform through static CA assessments in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Zeiler, MD PhD FRCSC, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre (HSC), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No